CLINICAL TRIAL: NCT03908853
Title: Pain Phenotyping of Patients With Bone Cancer Pain
Acronym: BonemetPAIN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Copenhagen (Other)
Collaborators: The Novo Nordic Foundation (Other)
Responsible Party: Principal Investigator, Anne-Marie Heegaard, Associate Professor, University of Copenhagen
Other Study IDs: H-18041465
Record Dates: First submitted 2019-03-28; First posted 2019-04-09 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-03

CONDITIONS: Pain; Bone Metastases; Metastatic Breast Cancer
MeSH Terms: conditions — Pain; Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Subjects with painful bone metastases caused by primary breast cancer.
- Controls: Gender and age matched healthy volunteers.

SUMMARY:
The study aims to describe and quantify pain related to metastatic bone disease. The study will include 50 subjects with disseminated breast cancer and 20 healthy subjects. The pain will be described and quantified through (1) pain specific questionnaires, (2) quantitative sensory testing that assess sensory changes to cold, heat and mechanical stimulation of the skin overlying the metastatic site, and (3) conditioned pain modulation that investigates impairment of the endogenous inhibitory pain pathway in humans.

DETAILED DESCRIPTION:
Cancer patients in palliative care point to pain as their most important and most feared symptom. Bone metastases are a common cause of cancer pain, and the patients are prone to transient severe pain exacerbations (breakthrough pain), which can occur spontaneously or be triggered by movement. Patients with bone metastases experience pain of such high intensity, that it affects not only physical activity, but also sleep, mood and social relations. This results in poor quality of life for the patients and poses an increasing clinical and socio-economical problem. The pain is difficult to treat and often requires high opioid doses which results in unacceptable adverse effects, and there is an unmet need of novel therapeutic options and treatment strategies.

Animal models of cancer-induced bone pain have suggested that pain arising from metastatic bone disease involve neuropathic and nociceptive pain mechanisms and, importantly, mechanisms that are specific to cancer-induced bone pain. Significant neuronal sprouting can occur at the metastatic site, and the inherent pain control system is found altered in animal models of cancer-induced bone pain; a system that can be exploited for treatment strategies and in the development of new analgesia. Yet, it is not known how the pre-clinical findings translate to patients.

Quantitative sensory testing is a psychophysical method that uses a battery of sensory stimuli with predetermined physical properties, thus allowing the capture and quantification of stimulus-evoked negative and positive sensory phenomena in humans. Conditioned pain modulation is a psychophysical experimental measure of the endogenous pain inhibitory pathway in humans, which can be used to detect an impairment of the descending inhibitory pain pathway.

This study aims to perform pain phenotyping of patients suffering from cancer-induced bone pain, through pain specific questionnaires, quantitative sensory testing and conditioned pain modulation.

ELIGIBILITY:
Inclusion Criteria:

* Woman
* Primary breast cancer
* Bone metastases
* Competent

Exclusion Criteria:

* Not fluent in spoken Danish
* Chemotherapy or radiation within the last 3 months
* Other chronic pain disease that may affect the quantitative sensory testing or conditioned pain modulation
* Alcohol or medicine abuse
* Pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 50 subjects with bone metastases caused by primary breast cancer and 20 healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2019-02-05 (Actual); Primary Completion 2022-02-01 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
Conditioned pain modulation (CPM) determined by cuff pressure algometry | 1 day
  CPM will be determined by placing two inflatable cuffs around the lower legs; one providing a test stimulus and the other a conditioning stimulus. First, the pressure pain detection and tolerance thresholds (kPa) are determined on each lower leg using an increasing pressure of 1 kPa/s; next a constant conditioning stimulus is applied to the dominant lower leg and 10 seconds later the pain pressure detection and tolerance threshold (kPa) are simultaneously determined on the non-dominant leg. The CPM effect is assessed as the percent difference between the measured thresholds on the non-dominant lower leg.
Sensory mapping with thermorollers and brush | 1 day
  Sensory changes to cold, warm and dynamic mechanical stimulation with thermo rollers (25°C and 40°C) and a standardized brush (No. 5, Somedic). Determination of area with either increased, decreased or painful changes.

SECONDARY OUTCOMES:
Mechanical pain threshold with PinPrick. | 1 day
  Determination of the mechanical pain threshold with PinPricks using a series of five ascending and five descending stimulus intensities (range 8 mN - 512 mN). The threshold is calculated as the geometric mean of the supra- and sub-threshold readings (mN).
Wind up ratio with Pin Prick | 1 day
  Determination of the pain rating (numeric rating scale, range 0-100) to 10 repeated stimuli with either a standardized brush or a PinPrick (256 mN). The wind up ratio is calculated as the arithmetic mean of the pain intensity rating for the series of stimuli divided by the arithmetic mean of the pain intensity rating for the single stimulus.
Cuff pressure pain threshold and pressure pain tolerance determined by cuff pressure algometry | 1 day
  Pressure pain detecting threshold and pain tolerance threshold (kPa) will be determined by placing two inflatable cuffs around the lower legs. The two thresholds are determined at the same time using an increasing pressure of 1 kPa/s.
Temporal summation of pressure pain | 1 day
  Determination of the pain rating (VAS, range 0-10) to 10 repeated stimuli with cuff pressure (pain tolerance threshold). The wind up ratio is calculated as the difference between the normalized mean of the pain intensity rating for the last series of stimuli divided by the normalized mean of the pain intensity rating for first stimuli.
Questionnaire - The Short Form Brief Pain Inventory | 1 day
  The short form Brief Pain Inventory measures pain intensity, localization of pain and influence on daily activities and quality of life through 9 items. All items cover the last 24 hours.
  Measurement of worst, least, average and current pain on a scale from 0-10, where 0 equals "no pain" and 10 equals "pain as bad as you can imagine"; the measures are used individually or combined into a mean severity score.
  Determination of pain localization using a pain drawing (human figure); the information is used qualitatively.
  Determination of pain relief on a scale from 0-100%. Measurement of how much pain interferes with daily activities, including general activity, walking, work, mood, enjoyment of life, relations with others, and sleep; the measurement is done on a scale from 0-10, where 0 equals "does no interference" and 10 equals "completely interferes"; the seven interference items are combined into a mean score.
Questionnaire - PainDETECT | 1 day
  Screens for neuropathic pain components through 13 items. Measurement of current, strongest and average pain within the last 4 weeks on a scale from 0-10, 0 equals "none" and 10 equals "maximal"; the measures are used individually.
  Marking of pain pattern (persistent, fluctuating) according to 4 pictures; a score from -1 to +1 is given depending on pain pattern.
  Determination of pain localization using a pain drawing and indication of pain radiating to other body regions; radiating pain will give a score of +2.
  Determination of the sensation of the pain (e.g. burning, prickling, numbness) using 7 items; the scale includes the following choices resulting in the indicated scores; never (0), hardly noticed (+1), slightly (+2), moderately (+3), strongly (+4), and very strongly (+5).
  The total score is calculated (ranging from 0-38) and the number used to determine the likelihood of a neuropathic pain component with 0-12 resulting in negative, 13-18 unclear and 19-30 positive.
Questionnaire - The Breakthrough Pain Questionnaire | 1 day
  The Breakthrough Pain Questionnaire is used to assess breakthrough pain intensity, frequency, duration, and triggering and relieving factors through 9 items. The obtained measures are used individually and some only qualitatively.
  Measurement of average background and breakthrough pain within the last 24 hours on a scale from 0-10, where 0 equals "no pain" and 10 equals "worst pain imaginable".
  Indication of breakthrough pain episodes within the last 24 hours. Indication of average duration of breakthrough pain episodes using six time intervals ranging from "less than one minute" to "more than 120 minutes"; indication of the time from onset to peak pain using five time intervals ranging from "less than 10 seconds" to "31-60 minutes"; and indication of the predictability of breakthrough pain episodes ranging from "never" to "always".
  Indication of triggering and relieving factors choosing statements such as "when I move", "when I sit" and "taking prescribed pain medication".
Questionnaire - Pain Catastrophizing Scale | 1 day
  The Pain Catastrophizing Scale assess catastrophising related to pain experience through 13 items.
  The subject evaluates 13 statements describing thoughts and feelings that may be associated to pain, e.g. "I feel I can't go on" and "I keep thinking of other painful events", and indicates the degree to which she has these thoughts when experiencing pain. The scale for all items includes the following choices resulting in the scores indicated in brackets; not at all (0), to a slight degree (+1), to a moderate degree (+2), to a great degree (+3), and all the time (+4).
  The total score is calculated (ranging from 0-52) with a score of 30 or more representing a clinically relevant level of catastrophizing. Three subscales can be calculated: rumination (sum of four items), magnification (sum of three items), and helplessness (sum of six items), with cut-off scores of for clinically relevant levels at 11, 5 and 13, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Marie Heegaard, PhD, Principal Investigator — University of Copenhagen
Locations (2):
- Denmark (2):
  - Department of Oncology, Rigshospitalet, Copenhagen
  - The Department of Oncology, Herlev Hospital, Herlev

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stromgren AS, Sjogren P, Goldschmidt D, Petersen MA, Pedersen L, Groenvold M. Symptom priority and course of symptomatology in specialized palliative care. J Pain Symptom Manage. 2006 Mar;31(3):199-206. doi: 10.1016/j.jpainsymman.2005.07.007. PMID 16563314
- [Background] Banning A, Sjogren P, Henriksen H. Treatment outcome in a multidisciplinary cancer pain clinic. Pain. 1991 Nov;47(2):129-134. doi: 10.1016/0304-3959(91)90195-4. No abstract available. PMID 1762805
- [Background] Mercadante S. Managing difficult pain conditions in the cancer patient. Curr Pain Headache Rep. 2014 Feb;18(2):395. doi: 10.1007/s11916-013-0395-y. PMID 24407750
- [Background] Laird BJ, Walley J, Murray GD, Clausen E, Colvin LA, Fallon MT. Characterization of cancer-induced bone pain: an exploratory study. Support Care Cancer. 2011 Sep;19(9):1393-401. doi: 10.1007/s00520-010-0961-3. Epub 2010 Aug 1. PMID 20680354
- [Background] Hald A, Nedergaard S, Hansen RR, Ding M, Heegaard AM. Differential activation of spinal cord glial cells in murine models of neuropathic and cancer pain. Eur J Pain. 2009 Feb;13(2):138-45. doi: 10.1016/j.ejpain.2008.03.014. Epub 2008 May 21. PMID 18499488
- [Background] Bloom AP, Jimenez-Andrade JM, Taylor RN, Castaneda-Corral G, Kaczmarska MJ, Freeman KT, Coughlin KA, Ghilardi JR, Kuskowski MA, Mantyh PW. Breast cancer-induced bone remodeling, skeletal pain, and sprouting of sensory nerve fibers. J Pain. 2011 Jun;12(6):698-711. doi: 10.1016/j.jpain.2010.12.016. Epub 2011 Apr 15. PMID 21497141
- [Background] Donovan-Rodriguez T, Urch CE, Dickenson AH. Evidence of a role for descending serotonergic facilitation in a rat model of cancer-induced bone pain. Neurosci Lett. 2006 Jan 30;393(2-3):237-42. doi: 10.1016/j.neulet.2005.09.073. Epub 2005 Oct 25. PMID 16256273
- [Background] Honore P, Rogers SD, Schwei MJ, Salak-Johnson JL, Luger NM, Sabino MC, Clohisy DR, Mantyh PW. Murine models of inflammatory, neuropathic and cancer pain each generates a unique set of neurochemical changes in the spinal cord and sensory neurons. Neuroscience. 2000;98(3):585-98. doi: 10.1016/s0306-4522(00)00110-x. PMID 10869852
- [Background] Falk S, Patel R, Heegaard A, Mercadante S, Dickenson AH. Spinal neuronal correlates of tapentadol analgesia in cancer pain: a back-translational approach. Eur J Pain. 2015 Feb;19(2):152-8. doi: 10.1002/ejp.530. Epub 2014 Jun 11. PMID 24917026
- [Background] Kennedy DL, Kemp HI, Ridout D, Yarnitsky D, Rice ASC. Reliability of conditioned pain modulation: a systematic review. Pain. 2016 Nov;157(11):2410-2419. doi: 10.1097/j.pain.0000000000000689. PMID 27559835
- [Background] Rolke R, Magerl W, Campbell KA, Schalber C, Caspari S, Birklein F, Treede RD. Quantitative sensory testing: a comprehensive protocol for clinical trials. Eur J Pain. 2006 Jan;10(1):77-88. doi: 10.1016/j.ejpain.2005.02.003. PMID 16291301
- [Background] Yarnitsky D, Granot M, Nahman-Averbuch H, Khamaisi M, Granovsky Y. Conditioned pain modulation predicts duloxetine efficacy in painful diabetic neuropathy. Pain. 2012 Jun;153(6):1193-1198. doi: 10.1016/j.pain.2012.02.021. Epub 2012 Apr 3. PMID 22480803